CLINICAL TRIAL: NCT02332135
Title: The Efficacy and Safety of Microwave Ablation for Mild-to-moderate Secondary Hyperparathyroidism Patients Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenhu Liu (Other)
Responsible Party: Sponsor-Investigator, Wenhu Liu, Professor, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJFH-EC/2014-101
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Secondary Hyperparathyroidism; Maintenance Hemodialysis
Keywords: microwave ablation; maintenance hemodialysis; mild-to-moderate Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- microwave ablation group (Experimental): patients in ultrasonic ablation will be treated by ultrasound guided percutaneous parathyroid gland microwave ablation
  Interventions: Procedure: microwave ablation
- control group (Active Comparator): patients in control group will be treated by active vitamin D and other general treatments according to the suggestions in K/DOQI guidelines
  Interventions: Drug: active vitamin D

INTERVENTIONS:
Procedure: microwave ablation — First, the investigators detect the iPTH levels of all the patients in the investigators' blood purification center. The patients whose iPTH are between 300pg/ml and 800pg/ml and who have parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan are chosen to involve in this study. Patients are divided into 2 groups at random, the control group and the microwave ablation group. In the microwave ablation group, patients will accept microwave ablation. Oral medicines, if needed, will be taken according to the the suggestions in K/DOQI guideline.
  Arms: microwave ablation group
Drug: active vitamin D — The control group will be treated by active vitamin D and other general treatment,such as dietary phosphate restriction and phosphate binders,according to the suggestions in K/DOQI guideline.
  Arms: control group

SUMMARY:
Microwave ablation, as a new method to therapy secondary hyperparathyroidism(SHPT), now is developing rapidly. However, it is still unknown whether it is effective to accept microwave ablation for hemodialysis patients with mild-to-moderate SHPT. In this prospective, randomised control and paried clinical trial study, the investigators will observe the efficiency and safety of microwave ablation in hemodialysis patients with mild-to-moderate secondary hyperparathyroidism. The patients in age-matched control group will accept active Vitamin D therapy.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism(SHPT) is common in hemodialysis(HD) patients. SHPT can damage cardiovascular system , bone system, and so forth. The treatment of SHPT of HD patients includes dietary phosphate restriction, the use of medicines, parathyroidectomy, and microwave ablation, which is a new method booming over the past decade. However, In the mainland of China, medical therapy is not always successful in achieving adequate control of SHPT. Oral medications have limitations as well as side effects. The patients may suffer from the injury of operation, hypoparathyroidism, or recurrence of hyperparathyroidism after parathyroidectomy. Moreover, the fear of operation for patients also limits its development. Thus, microwave ablation may become a valuable alternative treatment to help control SHPT in selected patients presenting with enlarged parathyroid gland(s) visible at ultrasonography. Nevertheless, nowadays there isn't a guideline for doctors to choose when to use microwave ablation to therapy SHPT. Furthermore, different experts have different views. Experts in Japan consider that, for SHPT , the earlier one takes microwave ablation, the better he may be, while others think, Just as parathyroidectomy, microwave ablation is merely used for the patient whose intact parathyroid hormone (iPTH) is more than 800pg/ml, or who has serious symptom. From their perspective, this is no proof that accepting microwave ablation for SHPT in early stage becomes better. However, as we all know, as the disease progresses, the therapy becomes increasingly difficult. Since microwave ablation is minimally invasive, safe,the investigators consider, patients who have parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan would get more benefit if they undergo microwave ablation the instant that SHPT is diagnosed. So, In this prospective, randomised control and paried clinical trial study, the investigators will observe the efficiency and safety of microwave ablation in hemodialysis patients with secondary hyperparathyroidism in early stage. First, the investigators detect the iPTH levels of all the patients in the investigators' blood purification center. The patients whose iPTH are between 300pg/ml and 800pg/ml and who have parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan are chosen to involve in this study. The patients with age-matched and iPTH between 300pg/ml and 800pg/ml were enrolled in this study. In the control group, patients will accept vitamin D to treat SHPT, according to the suggestions in K/DOQI guidelines. Meanwhile, in the microwave ablation group, patients will accept microwave ablation. Then, all of the patients will be followed for 24 months to compare the rate of achieving the target on iPTH level according to K/DOQI guidelines, the change of iPTH level after MWA,the rate of subjects developed into severe SHPT, as well as calcium and phosphorus level, Quality of Life and mortality in each group.

ELIGIBILITY:
Inclusion Criteria:

1. patients with age between 18-75 years.
2. patients with parathyroid nodular or diffuse hyperplasia demonstrated on ultrasound imaging or radioisotope scan.
3. patients in hemodialysis, whose iPTH is between 300pg/ml and 800pg/ml.

Exclusion Criteria:

1. primary or tertiary hyperparathyroidism(hyperparathyroidism after kidney transplantation).
2. patient who underwent total parathyroidectomy.
3. Known history of parathyroid or other neoplasias in the neck region.
4. History of neck trauma.
5. major surgery of neck in the last 3 months or in next 4months.
6. pregnant or lactating woman.
7. patients with severe liver disease and abnormal blood clotting mechanism.
8. patients with chronic wasting disease.
9. patients who is taking glucocorticoids.
10. patients who have other disorders affecting calcium and phosphorus metabolism.
11. patients whose concurrent illnesses,disability,or geographical residence would hamper attendance at required study visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Overall rate of achieving target for iPTH during the study period. | 12 months
  The blood level of intact iPTH will be detected every other month for stable patients.
The change of iPTH level after MWA. | 12 months
  The blood level of intact iPTH will be detected every other month for stable
The rate of subjects developed into severe SHPT | 12 months

SECONDARY OUTCOMES:
Calcitriol weekly dosage. | 12 months
  calcification score in every 6 months
Overall rate of achieving target for serum calcium and phosphorus. | 12 months
Changes of serum calcium and phosphorus after MWA. | 12 months
  The blood level of bone specific alkaline phosphatase will be detected every other months

CONTACTS AND LOCATIONS:
Overall Officials: Wenhu Liu, doctor, Study Chair — Beijing Friendship Hospital; Zongli Diao, master, Study Director — Beijing Friendship Hospital; Linxue Qian, doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friedship Hospital, Beijing, Beijing Municipality, China